CLINICAL TRIAL: NCT00821925
Title: Estimation of Osteoporosis' Prevalence in France: Pilot Study in the Department of the Alpes-Maritimes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 06-PP-04
Record Dates: First submitted 2009-01-12; First posted 2009-01-14 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2009-01

CONDITIONS: Osteoporosis
Keywords: osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: bone densitometry — All patients do a bone densitometry after the inclusion.

SUMMARY:
The purpose of this study is to estimate Osteoporosis' prevalence in France and is a pilot study in the Department of the Alpes-Maritimes.

ELIGIBILITY:
Inclusion Criteria:

* Patient member of Caisse Primaire d'Assurance Maladie

Exclusion Criteria:

* Patient incapable of understanding the questionary

Ages: 50 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2006-12

CONTACTS AND LOCATIONS:
Overall Officials: Liana Euller-Ziegler, PU-PH, Principal Investigator — Department of Rheumatology
Locations (1):
- Department of Rheumatology, Nice, France